CLINICAL TRIAL: NCT04474236
Title: Use of Lung Ultrasound for COVID-19 Patient's Initial Triage Assessment and Early Monitoring: a Pilot Study
Brief Title: Lung Ultrasound for COVID-19 Initial Triage and Monitoring
Acronym: QUICK
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0182; 2020-A01445-34 (Other: ID-RCB)
Record Dates: First submitted 2020-07-07; First posted 2020-07-16 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; Acute Respiratory Failure; Triage; Lung Ultrasound; CT Scan
Keywords: COVID-19; Acute Respiratory Failure; Triage; Lung Ultrasound; CT scan
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Adult (> 18 years) with Proven COVID-19 (specific PCR from respiratory track sample)
  Interventions: Other: thoracic lung ultrasound

INTERVENTIONS:
Other: thoracic lung ultrasound — Patients will be recruited the day of their hospital admission. All patients will be assessed by thoracic Computed Tomography scan then immediately before/after CT scan, patients will be clinically assessed (Q-SOFA, SpiO2/FiO2) and a lung ultrasound evaluation (mean time of evaluation 7 min +/- 3 min; fully respect of COVID-19 barrier measures) will be performed by an investigator. Patients clinical status and outcomes will be extracted from patient's medical file at day 1 and day 28 from patient's admission by investigators blinded from previously recorded lung ultrasound data.

SUMMARY:
The QUICK study main aim is to assess the predictive value at Day 1, of a model built on lung ultrasound (LUS) and clinical data, both recorded at hospital admission of COVID-19 patients.

DETAILED DESCRIPTION:
Initial triage assessment is the cornerstone of first-line medical management for COVID-19 patients. Only an accurate and fast evaluation of COVID-19 patients respiratory system integrity, can allow optimal treatment care and medical resources attribution. Despite its very large deployment, the use of thoracic Computed Tomography (CT scan) for COVID-19 patients severity assessment is currently debated. Actually CT-scan use in this setting: i) it is associated with risky in/out hospital patient's transport, both in terms of medical management of patient's critical conditions and risk of COVID-19 nosocomial transmission, ii) risks related to x-ray exposure iii) CT-scan is a snapshot of respiratory system integrity and does not provide data that might be used for patient's monitoring. LUS is a non-invasive, non-ionizing, fully bedside imaging tool. Investigators team has previously contributed to the development and validation of LUS for critically ill patient's management. To the extent of our knowledge, there is neither data regarding COVID-19 patient's LUS patterns, nor about the potential link between LUS data, patient's severity and outcome.

The investigators hypothesize that the combined use of LUS and clinical data (Q-SOFA score, SpiO2/FiO2) recorded at COVID-19 patients hospital admission, will allow to accurately predict short-term outcome. The investigators expect to predict at patient's hospital admission, the patient's clinical status at 24h: favorable (spontaneous ventilation with O2 < 6 l/min) or unfavorable (spontaneous ventilation with O2 > 6 l/min or under mechanical ventilation).

ELIGIBILITY:
Inclusion criteria:

* Adult (> 18 years).
* Proven COVID-19 (specific PCR from respiratory track sample)
* CT scan prescribed by physician in charge, independently of research.
* Patients consent (or surrogate decision maker's consent in case of need).

Exclusion criteria:

* Reduction or cessation of active treatment.
* Patient under guardianship, tutelage measure or judicial protection
* Patient deprived of liberty by judicial order
* No French health insurance.
* Pregnancy or nursing woman.
* Enrolled in another trial evaluating thoracic imaging.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pilot study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of a predictive model built on LUS and clinical (Q-SOFA, SpiO2/FiO2) data | Day 1
  Area Under the Curve (AUC) of a predictive model at 24h from hospital admission (Favorable vs Unfavorable), built on LUS (12 thoracic regions) and clinical (Q-SOFA, SpiO2/FiO2) data recorded at hospital admission.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of a predictive model built on CT scan and clinical (Q-SOFA, SpiO2/FiO2) data | Day 1
  Area Under the Curve (AUC) of a predictive model at 24h from hospital admission (Favorable vs Unfavorable), built on CT scan and clinical (Q-SOFA, SpiO2/FiO2) data recorded at hospital admission.
mortality | Day 28
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Benjamine SARTON, ph, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided